CLINICAL TRIAL: NCT07065552
Title: A Pre-Operative Window Study of Tirzepatide in Obesity-Driven Endometrial Cancer
Brief Title: Tirzepatide in Obesity-Driven Endometrial Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2415
Record Dates: First submitted 2025-06-04; First posted 2025-07-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Obesity
Keywords: tirzepatide; tumor microenvironment; insulin; lipid; mTOR signaling
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Insulin Resistance | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- endometrial carcinoma (Experimental): Obese women with endometrial carcinoma are included.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide will be administered once weekly, subcutaneously, and patients will be taught how to administer this drug at home. Patients will be started on a dose of 5 mg tirzepatide weekly for four weeks prior to surgical staging. .

SUMMARY:
LCCC2415 examines the antiproliferative effect of tirzepatide on the endometrium of endometrial cancer (EC). This is a pre-operative window clinical study. Endometrial biopsy samples from patients before tirzepatide treatment will be compared to their post-intervention hysterectomy specimens. If archival tissue is unavailable, a fresh biopsy will be taken before tirzepatide treatment. Post-intervention tissue will be collected from the hysterectomy specimen.

The hypothesis is that tirzepatide's anti-tumorigenic effects are due to both an improvement in the host's metabolic milieu (indirect effect) and a direct effect on the EC tumor microenvironment via the inter-related pathways of insulin, lipid, and mTOR signaling. Therefore, tirzepatide may be an innovative approach to effectively induce weight loss and inhibit tumor growth in EC, the most obesity-driven of all cancers.

DETAILED DESCRIPTION:
The primary objective is to determine if tirzepatide decreases proliferation in the tumors of EC patients. The effect of tirzepatide on the endometrium of 20 obese women with EC will be evaluated by comparing each patient's endometrial biopsy before tirzepatide treatment to their post-treatment hysterectomy specimen, through a pre- operative window study. These women will begin tirzepatide treatment for 4 weeks prior to standard-of-care (SOC) surgery. Subjects will have a single end-of-treatment visit 4 weeks after completing therapy and will be followed for 24 months via medical record abstraction to monitor weight loss maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of endometrioid histology cancer and scheduled to undergo hysterectomy and staging.
* Agree to comply with all required study assessments and visits including internet capabilities.
* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Age ≥ 18 at the time of consent.
* Body mass index of ≥30 kg/m2.
* Presumed clinically early-stage disease (disease confined to uterus only).
* ECOG ≤ 2 or Karnofsky Performance Status of > 50

Exclusion Criteria:

* Active infection requiring systemic therapy.
* Subject is pregnant or breast feeding.
* Taking any prescription medications or other drugs that may influence metabolism per discretion of investigator.
* Taking a central nervous system stimulant.
* Current psychological conditions that would be incompatible with participation in this study, as determined by investigator.
* Known sensitivities (i.e., urticaria and eczema) to GIP and GLP-1 receptor agonists.
* Have type 1 diabetes mellitus or latent autoimmune diabetes in adults or receiving treatment with insulin.
* Have a history of severe hypoglycemia or not be able to communicate an understanding of hypoglycemic symptoms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Proliferation | Baseline - Up to 6 weeks
  Change in Proliferation will be determined by immunohistochemical ( Ki-67 staining) analysis pre- (baseline) and post-tirzepatide treatment hysterectomy samples (at the time of surgery and end of treatment). The percentage of tumor cells that are positive for Ki-67, indicating they are in the active phases of the cell cycle (not resting). Low Ki-67 (<10-15%): Slower-growing tumor. Intermediate (15-30%): Moderately proliferative. High (>30%): Fast-growing, potentially more aggressive.

SECONDARY OUTCOMES:
Improvement in Diabetes | Baseline - Up to 6 weeks
  Diabetes status (yes/no) will be documented before and after tirzepatide treatment using the medical records and diabetes diagnostic criteria.
Improvement in HgbA1C level | Baseline - Up to 6 weeks
  HgbA1C level will be documented pre- and post-tirzepatide treatment.
Improvement in waist-to-hip ratio | Baseline - Up to 6 weeks
  The waist-to-hip ratio will be documented pre- and post-tirzepatide treatment.
Improvement in Body Mass Index | Baseline - Up to 6 weeks
  Body Mass Index (measured by dividing weight in kgs by height in meters) will be documented pre- and post-tirzepatide treatment.
Change in circulating levels of inflammatory cytokines | Baseline - Up to 6 weeks
  Serum levels of leptin, adiponectin, CRP, IL-1B, VEGFA, CCL3, IL-23, TNF-A, IL-6 pre- and post-tirzepatide treatment will be documented.
Change in sex hormones | Baseline - Up to 6 weeks
  Serum levels of estradiol, estrone, and sex hormone binding globulin pre- and post-tirzepatide treatment will be documented.
Change in Lipids | Baseline - Up to 6 weeks
  Serum levels of lipid panel pre- and post-tirzepatide treatment will be documented.
Change in insulin | Baseline - Up to 6 weeks
  Serum levels of fasting insulin pre- and post-tirzepatide treatment will be documented.
Change in Insulin-like Growth Factor 1 | Baseline - Up to 6 weeks
  Serum levels of Insulin-like Growth Factor 1 (IGF-1 ) pre- and post-tirzepatide treatment will be documented. IGF-1 is a hormone similar in structure to insulin and plays a crucial role in growth and development. Here are the key points about IGF-1:
Change in glucose | Baseline - Up to 6 weeks
  Serum glucose levels pre- and post-tirzepatide treatment will be documented.
Change in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), and Gamma-Glutamyl Transferase (GGT) levels | Baseline - Up to 6 weeks
  Serum liver function panel pre- and post-tirzepatide treatment will be documented. The same serum sample will be used to measure to determine Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), and Gamma-Glutamyl Transferase (GGT) levels. All participants will be analyzed using this single sample, and results will be reported in Units per Liter (U/L) for each enzyme.
Change in Apoptosis | Baseline - Up to 6 weeks
  Apoptosis will be assessed via immunohistochemistry before and after tirzepatide treatment.
Change in Ribonucleic Acid (RNA) sequence | Baseline - Up to 6 weeks
  RNA sequence will be assessed via immunohistochemistry in endometrial carcinoma specimen before and after tirzepatide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bae-Jump Victoria, MD PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials